CLINICAL TRIAL: NCT02707380
Title: The Effectiveness of Resistance Training on Glycemic Control for Patients With Type 2 Diabetes in Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-01994
Record Dates: First submitted 2016-02-22; First posted 2016-03-14 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes (T2DM); Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Resistance Training; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 Resistance Training Group (Active Comparator): Participants will perform 3 exercises, one of which will be a series of 7 muscle-strengthening exercises using body weight resistance and elastic resistance bands + 36 sessions of a standard cardiac rehabilitation program consisting of monitored exercise, nutritional guidance, and heart-healthy lifestyle education three times weekly.
  Interventions: Other: Resistance Training
- Group 2 Standard of Care (Active Comparator): Participants will perform 3 exercises that do not include the 7 muscle-strengthening exercises + 36 sessions of a standard cardiac rehabilitation program consisting of monitored exercise, nutritional guidance, and heart-healthy lifestyle education three times weekly.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Resistance Training — 7 muscle-strengthening exercises using body weight resistance and elastic resistance bands
  Arms: Group 1 Resistance Training Group
Other: Standard of Care — 3 exercises that do not include these 7 muscle-strengthening exercises
  Arms: Group 2 Standard of Care

SUMMARY:
This study is designed to investigate the effect of a structured resistance training program on glycemic control, measured by hemoglobin A1c (glycated hemoglobin), in patients with type 2 diabetes (T2DM) who are enrolled in outpatient cardiac rehabilitation. The investigator will compare the experimental group receiving resistance training to a control group made of patients enrolled in outpatient cardiac rehabilitation and perform 3 aerobic exercise modalities during their sessions, which is the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with T2DM and have been accepted for a standard outpatient cardiac rehabilitation program
* Cognitively able to comprehend the information presented in the program
* Cognitively able to give informed consent to participate in this study

Exclusion Criteria:

* Patients with orthopedic or neurological limitations that would prevent them from participating in the resistance training program or monitored exercise sessions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Comparison of Stress measured by change in heart rate | Baseline, One Year, 2 Years
Leg strength measured by assessing maximum weight subject can press one time on a leg press machine | up to 2 years
Paired T-test to compare test-retest Perceived exertion | up to 2 years
Paired T-test to compare test-retest Perceived dyspnea | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Francois Haas, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States